CLINICAL TRIAL: NCT03310242
Title: Comparison of Sunlight Exposure and Oral Vitamin D Supplementation on Serum 25-hydroxyvitamin D Concentration and Metabolic Markers in Korean Young Adults: a Randomized Clinical Trial
Brief Title: Comparison of Sunlight Exposure and Vitamin D Supplementation on Serum 25-hydroxyvitamin D Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H-1504-112-668
Record Dates: First submitted 2017-07-31; First posted 2017-10-16 (Actual); Last update posted 2017-10-31 (Actual); Status verified 2016-06

CONDITIONS: Vitamin D Deficiency; Cardiometabolic Risk Factors
MeSH Terms: conditions — Vitamin D Deficiency

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sunlight Exposure (Experimental): Everyday sunlight exposure around noon for 20-30 minutes for 8 weeks
  Interventions: Behavioral: Sunlight Exposure
- Vitamin D Supplementation (Experimental): Supplementation of vitamin D3 500 IU/day for 8 weeks
  Interventions: Dietary Supplement: Vitamin D Supplementation
- Placebo (Placebo Comparator): Intake of placebo for 8 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Behavioral: Sunlight Exposure — * Everyday sunlight exposure around noon for 20-30 minutes for 8 weeks
  * Completing a Sun Diary after sunlight exposure
  Arms: Sunlight Exposure
Dietary Supplement: Vitamin D Supplementation — - Supplementation of vitamin D3 500 IU/day for 8 weeks
  Arms: Vitamin D Supplementation
Other: Placebo — - Intake of placebo for 8 weeks
  Arms: Placebo

SUMMARY:
This study aimed to compare the effects between sunlight exposure and oral vitamin D supplementation on serum 25-hydroxyvitamin D concentration and metabolic markers in Korean young adults.

ELIGIBILITY:
Inclusion Criteria:

* Serum 25(OH)vitamin D < 12ng/mL
* age between 18 and 39 years
* Korean men and women

Exclusion Criteria:

* Vitamin D supplementation within 2 months
* Photosensitivity or UV allergy
* History of hyperparathyroidism/hypercalciuria/kidney stone/skin cancer and other cancer
* Under medication for hypertension, dyslipidemia, and diabetes
* Intake of photosensitive medicine during study period
* Exposure of strong UV (e.g., beach, sun tanning) during study period
* Pregnant/breast-feeding women

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2015-11-25 (Actual); Study Completion 2015-11-30 (Actual)

PRIMARY OUTCOMES:
Serum 25(OH)D | Baseline, 4 week, and 8 week
  Changes in serum 25(OH)D levels in ng/mL

SECONDARY OUTCOMES:
BMI | Baseline, 4 week, and 8 week
  Weight and height will be combined to report BMI in kg/m^2
Systolic blood pressure | Baseline, 4 week, and 8 week
  Systolic blood pressure changes in mmHg
Diastolic blood pressure | Baseline, 4 week, and 8 week
  Diastolic blood pressure changes in mmHg
Lipid panel | Baseline and 8 week
  Serum total cholesterol, triglycerides, HDL cholesterol, and LDL cholesterol in mg/dL
Fasting glucose | Baseline and 8 week
  Serum fasting glucose in mg/dL
AST | Baseline and 8 week
  Serum AST levels in mg/dL
ALT | Baseline and 8 week
  Serum ALT levels in mg/dL
GGT | Baseline and 8 week
  Serum AST, ALT, and GGT levels in mg/dL
Intact PTH | Baseline and 8 week
  Serum intact PTH levels in mg/dL
Whole body BMD and BMC | Baseline and 8 week
  Whole body BMD (g/cm^2) and BMC (kg) measured by DEXA
Lean body mass, fat mass, and percent fat | Baseline and 8 week
  Lean body mass (kg), fat mass (kg), and percent fat (%) measured by DEXA
Lean body mass, muscle mass, skeletal muscle mass, fat mass, and percent fat | Baseline, 4 week, and 8 week
  Lean body mass (kg), muscle mass (kg), skeletal muscle mass (kg), fat mass (kg), and percent fat (%) measured by body impedance analysis
EQ-5D-5L | Baseline, 4 week, and 8 week
  Quality of life measured using EQ-5D-5L scale. The EQ-5D is a standardised measure of health status developed by the EuroQol Group in order to provide a simple, generic measure of health status. In description part, health status is measured in terms of five dimensions (5D); mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The respondents self-rate their level of severity for each dimension using three-level (EQ-5D-3L) or five-level (EQ-5D-5L) scale. The 5-level version of EQ-5D (EQ-5D-5L) was developed to improve such constraints of the three-level scale.
  EQ-5D-5L scale can define 3,125 (=5^5) different health states, and the 5-digit number can be converted into a preference weight which is also referred to as a single weighted index score. The index score of a value set derived from the general population sample can be regarded as a "societal valuation of the respondent's health state" in that country.

CONTACTS AND LOCATIONS:
Overall Officials: Hee-Kyung Joh, PhD, Principal Investigator — Seoul National University College of Medicine/Seoul National University Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Joh HK, Hwang SS, Cho B, Lim CS, Jung SE. Effect of sun exposure versus oral vitamin D supplementation on serum 25-hydroxyvitamin D concentrations in young adults: A randomized clinical trial. Clin Nutr. 2020 Mar;39(3):727-736. doi: 10.1016/j.clnu.2019.03.021. Epub 2019 Mar 21. PMID 30987813